CLINICAL TRIAL: NCT00002384
Title: Vistide (Cidofovir Intravenous) Treatment IND Protocol for Relapsing Cytomegalovirus Retinitis in Patients With AIDS
Brief Title: A Study of Cidofovir in the Treatment of Cytomegalovirus (CMV) of the Eyes in Patients With AIDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gilead Sciences (Industry)
Collaborators: Anderson Clinical Research (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 276A; GS-95-120; 96ACR-GIL1
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-08

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections | interventions — Cidofovir

INTERVENTIONS:
Drug: Cidofovir

SUMMARY:
Incomplete Closed Protocol

ELIGIBILITY:
Information not available

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

REFERENCES:
- [Background] Stagg RJ, Gathe J, Lieberman RM, Nuessle SJ, Davis JL, Ruane P, Bellman PC, Horgan M, Jaffe HS. The Vistide (cidofovir injection) treatment IND for relapsing CMV retinitis (CMV-R). Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:120 (abstract no 306)